CLINICAL TRIAL: NCT06048627
Title: Clinical Investigation to Assess the Efficacy of an Antimicrobial Mouthrinse in the Reduction of Established Plaque and Gingivitis: a 6-month Clinical Study
Brief Title: Anti-gingivitis Mouthrinse
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-2022-10-MER-MW-JG
Record Dates: First submitted 2023-09-16; First posted 2023-09-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-04

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mouthwash Test (Active Comparator)
  Interventions: Drug: Amine/zinc lactate/fluoride system
- Mouthwash Experimental (Experimental)
  Interventions: Drug: negative control

INTERVENTIONS:
Drug: Amine/zinc lactate/fluoride system — Amine/zinc lactate/fluoride system (250 ppm F), meridol®, Colgate-Palmolive
  Arms: Mouthwash Test
Drug: negative control — Sodium fluoride mouthwash 250 ppm
  Arms: Mouthwash Experimental

SUMMARY:
The purpose of this study is to prove whether a fluoride/zinc lactate containing mouthrinse is able to reduce dental plaque and gingival inflammation in patients who have gingivitis when applied twice daily during brushing at home over a period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Availability for the six-month duration of the clinical research study.
* Good general health.
* Minimum of 20 uncrowned permanent natural teeth (excluding third molars).
* Initial gingivitis index of at least 1.5 as determined by the use of the Gingival Index (Löe 1967).
* Initial plaque index of at least 1.5 as determined by the use of the Plaque Index (Turesky et al. 1970).
* Signed Informed Consent Form.

Exclusion Criteria:

* Presence of orthodontic bands.
* Malign tumor(s) of the soft or hard tissues of the oral cavity.
* Antibiotic use any time during the one-month period prior to entry into the study.
* Participation in any other clinical study or test panel within the one month prior to entry into the study.
* Dental prophylaxis during the past two weeks prior to baseline examinations.
* History of allergies to oral care/personal care consumer products or their ingredients.
* On any prescription medicines that might interfere with the study outcome.
* An existing medical condition that prohibits eating or drinking for periods up to 4 hours.
* History of alcohol or drug abuse.
* Self-reported pregnant or lactating subjects.
* Participants who have systemic diseases that require regular systemic medication intake that may affect the gingival condition (e.g. antibiotics, phenytoin, nifedipine, cyclosporine, steroids, antiphlogistics).
* Participants who require antibiotic treatments for dental appointments.
* Participants with current moderate or severe chronic or aggressive periodontitis (periodontitis screening index [PSI] >2 in more than 2 sextants or PSI >3).
* Subjects with caries requiring treatment (e.g., caries with cavity) or other oral diseases (including gingival hyperplasia, diseases of the oral mucosa);
* Smokers or/and users of tobacco products.
* Persons, who are unable to give their consent (e.g., persons who have limited legal capacity)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Whole-mouth Mean Modified Gingival Index (MGI) | Baseline, 3 weeks, 12 weeks, 24 weeks
  Gingivitis, gingival severity and gingival, interproximal scores as measured by the Gingival Index as difference from baseline to 24 weeks between the study groups.

SECONDARY OUTCOMES:
Turesky Modification of the Quigley Hein Plaque Index (PI) | Baseline, 3 weeks, 12 weeks, 24 weeks
  Plaque, plaque severity and plaque interproximal scores as measured by the Plaque Index as difference from baseline to 24 weeks between the study groups and at each time-point.
Intraoral scans | Baseline, 3 weeks, 12 weeks, 24 weeks
  Quantitative changes & before/after imagery from intraoral scans
Patient-reported experiences | Baseline, 3 weeks, 12 weeks, 24 weeks
  Changes in participant-reported experience as determined through participant-questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Technische Universität Dresden, Dresden, Germany

IPD SHARING:
Plan to Share IPD: No